CLINICAL TRIAL: NCT04603703
Title: Effects of Thrust Joint Manipulation of Sacroiliac Joint in Chronic Piriformis Syndrome
Brief Title: Sacroiliac Joint Manipulation Effect in Chronic Piriformis Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00693 Benish Shahzadi
Record Dates: First submitted 2020-10-13; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Piriformis Syndrome
Keywords: High Velocity Low Amplitude Thrust; Piriformis Syndrome; Sacroiliac joint manipulation
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Both groups were treated simultaneously with their specified treatment techniques within given duration.
Who Masked: Participant
Masking Description: Participants did not know which treatment techniques are given in the specified groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVLAT Manipulation (Experimental): Ultrasound, moist hot pack, piriformis stretching, myofascial release, gluteal muscles strengthening, sciatic neurodynamics, HVLAT
  Interventions: Other: HVLAT Manipulation
- Conventional physical therapy (Active Comparator): Ultrasound, moist hot pack, piriformis stretching, myofascial release, gluteal muscles strengthening, sciatic neurodynamics
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: HVLAT Manipulation — Ultrasound for 10 mins/1 set/ (3 days/ week), Moist hot pack for 10 mins/1 set/ (3 days/ week), Piriformis stretching for 7 sec hold/ 7 repititions/ 1 set/ (3 days/ week), Myofascial release of lumbosacral paraspinal muscles for 3 mins/ 1 set/ (3 days/ week), Gluteal muscles strengthening for 10 sec hold/ 5 reps/ 1 set/ (3 days/ week), Sciatic Neurodynamics with 10 oscillations/ 3 sets/(3 days/ week), HVLAT manipulation/ 1 rep/ 1set/ (3 days/ week),
  A total of 2 weeks (6 sessions, 3 sessions/ week) were given each consisting of 30 mins.
  Arms: HVLAT Manipulation
Other: Conventional Physical Therapy — Ultrasound for 10 mins/1 set/ (3 days/ week), Moist hot pack for 10 mins/1 set/ (3 days/ week), Piriformis stretching for 7 sec hold/ 7 repititions/ 1 set/ (3 days/ week), Myofascial release of lumbosacral paraspinal muscles for 3 mins/ 1 set/ (3 days/ week), Gluteal muscles strengthening for 10 sec hold/ 5 reps/ 1 set/ (3 days/ week), Sciatic Neurodynamics with 10 oscillations/ 3 sets/(3 days/ week),
  A total of 2 weeks (6 sessions, 3 sessions/ week) were given each consisting of 30 mins.
  Arms: Conventional physical therapy

SUMMARY:
The objective of the study was to determine the effects of sacroiliac joint thrust manipulation on pain, pain pressure threshold, piriformis length and straight leg raise, in chronic piriformis syndrome.

DETAILED DESCRIPTION:
In 2017, a systematic review was conducted to measure the effectiveness of physical therapy approach for relieving the SIJ pain linked with PS. Participants were administered with conservative physical therapy, Kinesiology taping and sacroiliac joint manipulation in group A, group B and group C respectively. They have concluded that Sacroiliac joint manipulation was more effective as compare to the rest of the physiotherapy approach in lowering the SIJ pain associated with piriformis syndrome.

In 2014, an experimental study was conducted to compare the effects of nerve mobilization technique with conventional physical therapy approach. Pre and post treatment data was taken from the respective participants. The results of this study concluded that there is a significant differences in the outcome measures of both groups and nerve MOBS were proven to be more effective in relieving the sciatic nerve radiating pain associated with inflamed piriformis muscle in PS.

A study in July, 2012 was conducted to compare the effects of two possible physical therapy treatments in lowering the low back pain threshold associated with piriformis syndrome. These two techniques were METs and SCS. Their results concluded that both Muscle energy technique and Strain counter strain were proved to be equally effective in the management of functional disability and pain in low back associated with chronic PS.

An RCT was conducted in 2011, to measure the effectiveness of two possible manipulation methods which can be applied in patients with chronic piriformis syndrome. According to this study, manipulating the of SIJ along with lumber manipulation is more effective as compare to the SIJ manipulation alone to regain the total piriformis length for patients with Chronic PS.

Another study was conducted by Gopal Nambi and colleagues in Saudi Arabia. It was concluded that Program comprises of Post Isometric Relaxation is more effective as compare to conservative physical therapy in alleviating the pain, improving hip ROM and functional improvement in participants with PS.

ELIGIBILITY:
Inclusion Criteria:

* Patients having alteast 3 months chronic Piriformis syndrome
* FAIR test positive
* Unilateral or bilateral Piriformis Syndrome

Exclusion Criteria:

* Lumber Prolapsed Intervertebral Disc (PIVD)
* Patients having hip osteoarthritis
* Sacroiliatis (FABER test, Mennell's test, Sacral Thrust Test, Compression test, Distraction test, thigh thrust test)
* Lumbosacral instability
* Patients having any joint replacement in lumbosacral and hip regions.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6th Day
  Changes from baseline, Numeric Pain Rating Scale is a scale for pain starting from 0 to 10 where 0 indicates no pain and 10 indicates severe pain.

SECONDARY OUTCOMES:
Pressure Pain Threshold | 6th Day
  Changes from baseline, pressure pain Threshold were taken with the help of Algometer.
Piriformis Length | 6th Day
  Changes from the baseline, Piriformis Length were taken with the help of Goniometer.
Straight Leg Raise | 6th Day
  Changes from baseline, Straight Leg Raise were taken with the help of Inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, Phd, Principal Investigator — Riphah International University
Locations (1):
- Max Rehab & Physical Therapy Centre G-8 Markaz, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Subahi M, Alayat M, Alshehri MA, Helal O, Alhasan H, Alalawi A, Takrouni A, Alfaqeh A. The effectiveness of physiotherapy interventions for sacroiliac joint dysfunction: a systematic review. J Phys Ther Sci. 2017 Sep;29(9):1689-1694. doi: 10.1589/jpts.29.1689. Epub 2017 Sep 15. PMID 28932014
- [Background] Kutty RK, Gebrekidan HG, Lerebo WT, Gebretsadik MA. Neural mobilization a therapeutic efficacy in a piriformis syndrome model: an experimental study. International journal of physiotherapy and research. 2014;2(3):577-83.
- [Background] Ellythy MA. Efficacy of muscle energy technique versus strain counter strain on low back dysfunction. Bulletin of Faculty of Physical Therapy. 2012;17(2).
- [Background] Rodrigue T, Hardy RW. Diagnosis and treatment of piriformis syndrome. Neurosurg Clin N Am. 2001 Apr;12(2):311-9. PMID 11525209
- [Background] Bose GNSC, Dusad G. EFFECT OF RECIPROCAL INHIBITION AND POST ISOMETRIC RELAXATION; TYPES OF MUSCLE ENERGY TECHNIQUE IN PIRIFORMIS SYNDROME-A COMPARATIVE STUDY.